CLINICAL TRIAL: NCT06868160
Title: Neurotech PD Gait: Multisite Non-invasive Electrical Stimulation to Optimize Motor-cognitive Rehabilitation Response in Parkinson's Disease Subjects With Postural Instability and Gait Disorders
Brief Title: Comparison of Different Non-invasive Electrical Stimulation Protocols to Facilitate Rehabilitation in Parkinson's Disease Subjects With Postural Instability and Gait Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Prof., IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NEUROTECH_001 PD gait
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Gait; Rehabilitation; Biomarkers; Magnetic Resonance Imaging; Functional Near Infrared Spectroscopy; Non-invasive Electrical Stimulation; Electroencephalogram
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Every patient will undergo two rounds of training (6 weeks) with a 8-week washout period in between. Patients will be randomized in two parallel groups: 1/3 of the patients will receive two rounds of rehabilitation + SHAM stimulation; 2/3 of the patients will receive two rounds of rehabilitation + non-invasive STIMULATION.
  Patients in the STIMULATION group will be further randomized in two groups both receiving tDCS stimulation combined with tsDCS or SHAMtsDCS in a crossover design: one group will receive a first round of rehabilitation + tDCS + tsDCS followed by a round of rehabilitation + tDCS + SHAM tsDCS; the other group will receive the same treatment in an inverted order.
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessor blinded will be neurologists, neuropsychologists and physiotherapists who will perform the evaluations at each time point.
  Patients will not know if they are receiving sham or real stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- REHAB+SHAM (Active Comparator): Dual-task gait/balance training consisting of action observation training (AOT) and motor imagery (MI) combined with practicing the observed-imagined exercises. Patients will receive SHAM stimulation.
  Interventions: Behavioral: Rehabilitation; Device: SHAM tDCS; Device: SHAM tsDCS
- REHAB+tDCS+tsDCS (Experimental): Patients will perform the same exercises as REHAB+SHAM group, combined with non-invasive stimulation. Non-invasive stimulation will be administered using tDCS (DorsoLateral Prefrontal Cortex) combined with tsDCS for the first cycle (6 weeks). During the second cycle (6 weeks after 8-week washout) patients will receive tDCS + sham tsDCS.
  Interventions: Behavioral: Rehabilitation; Device: tDCS; Device: tsDCS (first cycle); Device: SHAM tsDCS (second cycle)
- REHAB+tDCS+SHAMtsDCS (Active Comparator): Patients will perform the same exercises as REHAB+SHAM group, combined with non-invasive stimulation. Non-invasive stimulation will be administered using tDCS (DorsoLateral Prefrontal Cortex) combined with SHAM tsDCS for the first cycle (6 weeks). During the second cycle (6 weeks after 8-week washout) patients will receive tDCS + tsDCS.
  Interventions: Behavioral: Rehabilitation; Device: tDCS; Device: tsDCS (second cycle); Device: SHAM tsDCS (first cycle)
- Healthy subjects (No Intervention): Age- and sex-matched healthy subjects recruited to compare gait, neuropsychological, serum, functional magnetic resonance imaging and neurophysiological characteristics at baseline

INTERVENTIONS:
Behavioral: Rehabilitation — Two cycles of dual-task gait/balance training consisting of action observation training (AOT) and motor imagery (MI) combined with practicing the observed-imagined exercises.
  Three 1-hour sessions per week for 6 weeks. Cycle repeated after 8-week washout period.
  Arms: REHAB+SHAM; REHAB+tDCS+SHAMtsDCS; REHAB+tDCS+tsDCS
Device: SHAM tDCS — SHAM stimulation will be performed using the same montage used for transcranial and spinal stimulation, however an initial current is delivered and programmed to fade off in a brief period of time.
  Arms: REHAB+SHAM
Device: tDCS — Anodic tDCS with the anode placed on the of the left DorsoLateral Prefrontal Cortex. Patients will undergo 30 minutes tDCS session preceding rehabilitation
  Arms: REHAB+tDCS+SHAMtsDCS; REHAB+tDCS+tsDCS
Device: tsDCS (first cycle) — Anodic spinal cervical stimulation with anode electrode placed on the spinous process of C3 vertebra and cathode placed on T3. Patients will undergo 30 minutes stimulation session preceding rehabilitation during the first cycle (6 weeks)
  Arms: REHAB+tDCS+tsDCS
Device: tsDCS (second cycle) — Anodic spinal cervical stimulation with anode electrode placed on the spinous process of C3 vertebra and cathode placed on T3. Patients will undergo 30 minutes stimulation session preceding rehabilitation during the second cycle (6 weeks after 8-week washout)
  Arms: REHAB+tDCS+SHAMtsDCS
Device: SHAM tsDCS (first cycle) — SHAM stimulation will have the same montage as tsDCS but run in SHAM more with an initial stimulation at standard intensity, followed by a programmed fade off after a brief time period. Patients will undergo 30 minutes of SHAM stimulation session preceding rehabilitation during the first cycle (6 weeks)
  Arms: REHAB+tDCS+SHAMtsDCS
Device: SHAM tsDCS (second cycle) — SHAM stimulation will have the same montage as tsDCS but run in SHAM more with an initial stimulation at standard intensity, followed by a programmed fade off after a brief time period. Patients will undergo 30 minutes of SHAM stimulation session preceding rehabilitation during the second cycle (6 weeks after 8-week washout)
  Arms: REHAB+tDCS+tsDCS
Device: SHAM tsDCS — SHAM stimulation will have the same montage as tsDCS but run in SHAM more with an initial stimulation at standard intensity, followed by a programmed fade off after a brief time period. Patients will undergo 30 minutes of SHAM stimulation session preceding rehabilitation
  Arms: REHAB+SHAM

SUMMARY:
The trial will include 51 adult participants with Parkinson's disease and postural instability and gait disorders (PD-PIGD) and 20 age- and sex-matched healthy controls.

At baseline (T0) patients will undergo neurological and cognitive/behavioural assessments, gait/balance evaluation, neuroimaging/neurophysiology assessments including brain magnetic resonance imaging (MRI), functional Near Infrared Spectroscopy (fNIRS) and Electroencephalography (EEG) acquisitions to assess brain activity, connectivity and structural changes, and blood sample.

PD-PIGD patients will be randomly allocated in two training groups: the REHAB+SHAM group and the REHAB + STIM group.

The REHAB+SHAM group will perform 2 cycles of dual-task gait/balance training consisting of action observation training (AOT) and motor imagery (MI) combined with practicing the observed-imagined exercises (an approach that has been demonstrated to be effective to improve gait and mobility in PD-PIGD), additionally they will undergo SHAM transcranial and trans-spinal stimulation. SHAM stimulation will be performed using the same montage used for transcranial and spinal stimulation (explained below), however an initial current is delivered and programmed to fade off in a brief period of time.

The REHAB + STIM group will perform the same exercises combined with non-invasive stimulation.

Non-invasive stimulation will be administered using tDCS with trans-spinal Direct Current Stimulation (tsDCS) or transcranial Direct Current Stimulation (tDCS) alone combined with SHAMtsDCS.

This design will aid in determining not only whether non-invasive stimulation can enhance rehabilitation outcomes but also whether the combination of tDCS and tsDCS could lead to improved results compared to tDCS alone.

The motor-cognitive training of the REHAB+SHAM group will consist of 2 cycles of SHAM stimulation and training lasting 6 weeks, 3 times per week, about 1 hour each session, separated by a 8-week washout period.

The REHAB + STIM group will undergo 2 cycles of the 6-week training, separated by a 8-week washout period with a cross-over design: half of subjects will first receive 6-week training with tDCS+SHAMtsDCS followed by 6-week tDCS+ tsDCS, while the other half will follow the reverse order, according to a randomization procedure.

After the training (i.e., 6-week visit [W6] and 20-week visit [W20]), PD-PIGD patients will be re-evaluated through neurological, cognitive/behavioural, gait/balance, neuroimaging/neurophysiology assessments and blood sample.

These measures (except for MRI at 14-week [W14] visit) will be also repeated at W14 and 28-week follow-up visits to assess maintenance of results.

20 healthy controls will also be recruited and evaluated at baseline. They will undergo the same assessments administered to PD-PIGD patients at T0 (neurological, cognitive/behavioural assessments, gait/balance evaluation using gait analysis systems, neuroimaging/neurophysiology, blood sample).

ELIGIBILITY:
Inclusion Criteria:

* 45 years < age ≤ 85 years
* Idiopathic PD according to the Movement Disorders Society (MDS) diagnostic criteria
* Hoehn & Yahr (H&Y) score ≤ 4
* PIGD phenotype
* Stable dopaminergic medication for at least 4 weeks and without any changes during the observation period (28 weeks)
* No dementia according to Litvan's criteria and Mini-Mental Status Examination score (MMSE) ≥ 24
* No significant tremor/involuntary movements that could determine artifacts during the MRI acquisition
* Oral and written informed consent to study participation

Healthy controls' inclusion criteria:

* Sex-matched and age-matched (age range: mean age of PD years ± 15 years)
* Oral and written informed consent to study participation

Exclusion Criteria:

* Any major systemic, psychiatric, neurological, visual, and musculoskeletal disturbances or other causes of walking inability
* Medical conditions or substance abuse that could interfere with cognition
* Pacemaker or other implanted neurostimulation devices in the head/neck district
* (Other) Contraindications to undergoing MRI examination
* Brain damage at routine MRI, including extensive cerebrovascular disorders
* Denied oral and written informed consent to study participation
* Significant scalp traumatic or surgical wounds or scalp alterations that could determine a risk of infection in the site of non-invasive stimulation or the spread of excessive current from the device (only for patients receiving the neurostimulation).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Total execution time of Timed Up and Go test with cognitive dual-task (TUG-COG) | Baseline, week 6, week 14, week 20 and week 28
  Changes in time taken to complete the timed up and go test with cognitive dual-task: patients are asked to stand up from a chair, walk for three meters, turn and walk back to the chair while counting backwards by 3 starting from 100. Assessment during ON medication phase

SECONDARY OUTCOMES:
Total execution time of Timed Up and Go test (TUG) | Baseline, week 6, week 14, week 20 and week 28
  Changes in time taken to complete the timed up and go test: patients are asked to stand up from a chair, walk for three meters, turn, and walk back to the chair. Assessment during ON medication phase
Total execution time of Timed Up and Go test with manual dual-task (TUG-MAN) | Baseline, week 6, week 14, week 20 and week 28
  Changes in time taken to complete the timed up and go test with manual dual-task: patients are asked to stand up from a chair, walk for three meters, turn, and walk back to the chair while holding a glass full of water. Assessment during ON medication phase
Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score | Baseline, week 6, week 14, week 20 and week 28
  MDS-UPDRS evaluates various aspects of Parkinson's disease including non-motor and motor experiences of daily living and motor complications. The MDS-UPDRS contains 65 items divided in four parts (Part I - "non-motor experiences of daily living", Part II - "motor experiences of daily living", Part III - "motor examination", Part IV - "motor complications. Each item is assessed with a 0 to 4 rating system. The total score ranges from 0 to 260 with higher score indicating more severe symptoms. Assessment during ON medication. Only part III assessed also without medication (OFF).
Brain functional changes during functional magnetic resonance imaging (MRI) tasks | Baseline, week 6, week 20 and week 28
  Changes in functional MRI brain activity assessed during a motor task, a cognitive task and a dual-task. Assessment during OFF medication phase, at least 12 hours after last medication assumption.
Changes at resting-state functional Near-Infrared Spectroscopy (fNIRS) | Baseline, week 6, week 14, week 20 and week 28
  Changes in the continuous spectral wave of brain resting activity
Changes in Electroencephalography (EEG) signal | Baseline, week 6, week 14, week 20 and week 28
  Changes in electrical brain activity during resting with eyes open and eyes closed
Serum concentration of Neurofilament light chain (NfL) | Baseline, week 6, week 14, week 20 and week 28
  Serum biomarker of neuroprotection/neurodegeneration
Activity Balance Confidence questionnaire (ABC) score | Baseline, week 6, week 14, week 20 and week 28
  This questionnaire assesses patient-referred balance confidence during 16 daily tasks. Subjects rate their confidence while doing each activity from 0 (no confidence) to 100 (full confidence). Assessment during ON medication phase.
10-meter walk test (10MWT) time | Baseline, week 6, week 14, week 20 and week 28
  Time taken to walk 10 straight meters. Test performed at comfortable and maximal speed. Assessment during ON medication phase.
Mini Balance Evaluation System Test (MiniBESTest) score | Baseline, week 6, week 14, week 20 and week 28
  Assessment of different balance systems (anticipatory, reactive postural control, sensory orientation, dynamic gait). MiniBESTest includes 14 items with a score from 0 (severe/unable) to 2 (normal). The maximum score is 28 and a higher score indicates a better balance. Assessment during ON medication phase.
Five-time sit-to-stand (5STS) time | Baseline, week 6, week 14, week 20 and week 28
  This test measures the amount of time it takes for a patient to stand up and sit down five times in a row, as quickly as possible with arms folded across their chest. Assessment during ON medication phase.
Parkinson's Disease Questionnaire (PDQ-39) score | Baseline, week 6, week 14, week 20 and week 28
  Parkinson's Disease Questionnaire investigates the quality of life of PD patients. It includes 39 questions with 5 possible answers (never, occasionally, sometimes, often, always) and 8 sub-items related to mobility, activities of daily living, emotional well-being, signs of discouragement, social support, cognitions, communication and bodily discomfort. The maximum score is 100 and a low score is an indicator of a good quality of life. Assessment during ON medication phase.
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | Baseline, week 6, week 14, week 20 and week 28
  This questionnaire assesses motor imagery abilities. The Kinesthetic and Visual Imagery Questionnaire (KVIQ) includes 10 items assessing the clarity of the image and the intensity of the sensations that the subject is able to imagine from the first-person perspective (both right and left sides) on a five-point ordinal scale. Total score ranges from 0 to 50 with higher score indicating better motor imagery abilities. Assessment during ON medication phase.
Vividness of Movement imagery Questionnaire (VMIQ) | Baseline, week 6, week 14, week 20 and week 28
  This questionnaire measures vividness of imagery in different visual imagery modalities (first and third person view) and kinaesthetic modality.
  Patients, for each imagery modality, give a score from 1 (best) to 5 (worse) to the clarity/intensity of 12 imagined actions.
Parkinson Fatigue Scale (PFS) | Baseline, week 6, week 14, week 20 and week 28
  Patient-rated scale that reflects the physical aspects of fatigue in patients with Parkinson's Disease (PD) and measures both the presence of fatigue and its impact on daily function
Fatigue Severity Scale (FSS) | Baseline, week 6, week 14, week 20 and week 28
  9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle
Modified Fatigue Impact Scale (M-FIS) | Baseline, week 6, week 14, week 20 and week 28
  Provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning
New Freezing of Gait Questionnaire (NFoG-Q) | Baseline, week 6, week 14, week 20 and week 28
  This is a self-reported questionnaire that measures freezing of gait. It consists of 9 items with a total score ranging from 0 (no freezing) to 28. Higher score indicates worse freezing. Assessment during ON medication phase.
Stride length | Baseline, week 6, week 14, week 20 and week 28
  Gait parameter obtained using wearable motion sensors. Assessment during ON medication phase.
Gait velocity | Baseline, week 6, week 14, week 20 and week 28
  Gait parameter obtained using wearable motion sensors. Assessment during ON medication phase.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, week 6, week 14, week 20 and week 28
  This battery of cognitive tests assesses executive functions, memory and visuospatial abilities. Each subtest of the CANTAB battery provides outcome measures in terms of accuracy (right answers, errors and/or missing answers) and reaction times (highest scores are worse) for every condition within the subtest (the different conditions present with different levels of cognitive load). Assessment during ON medication phase.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Neurotech Hub, Milan, Italy

IPD SHARING:
Plan to Share IPD: No